CLINICAL TRIAL: NCT06956430
Title: How Does Heat Stress Affect Telomere Length? A Pilot Randomized Controlled Trial in Urban Bangladesh
Brief Title: Mitigating Heat Stress Among Rickshaw Drivers in Bangladesh
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of California, Berkeley (Other)
Collaborators: International Centre for Diarrhoeal Disease Research, Bangladesh (Other); North South University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Single | Purpose: Prevention
Other Study IDs: 2023-05-16316
Record Dates: First submitted 2025-04-25; First posted 2025-05-04 (Actual); Last update posted 2025-05-21 (Actual); Status verified 2025-05

CONDITIONS: Core Temperature; Telomere Length, Mean Leukocyte; Kidney Function Issue
Keywords: heat stress; heat strain; rickshaw; heart rate; heart rate variability; sleep quality; Bangladesh
MeSH Terms: conditions — Heat Stress Disorders; Sleep Initiation and Maintenance Disorders

STUDY DESIGN:
Intervention Model Description: Stepped-wedge randomized controlled trial
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Manual rickshaw (No Intervention): Rickshaw drivers will use manually powered rickshaws
- Battery-powered rickshaw (Experimental): Rickshaw drivers will use battery-powered rickshaws
  Interventions: Device: Battery-powered rickshaw

INTERVENTIONS:
Device: Battery-powered rickshaw — A battery-powered rickshaw is a rickshaw where the wheels are turned by a small electric motors powered by a battery.
  Arms: Battery-powered rickshaw

SUMMARY:
The goal of the experimental study is to understand the impact of heat stress on core temperature and telomere length. Investigators will recruit rickshaw drivers who use manual power to push their rickshaws and randomly assign half of them to receive battery-powered rickshaws to use for four months. Investigators will assess how this change impacts their core body temperature while they work, the length of their telomeres (caps on the end of DNA that are associated with aging), and kidney function.

DETAILED DESCRIPTION:
Personal exposure to heat may be elevated above ambient temperatures if an individual is very active (which generates metabolic heat) or wears clothing that prevents cooling. Age can influence the consequences of heat stress. Older adults are at elevated risk of adverse impacts from heat stress due to their reduced ability to dissipate heat. Heat stress is particularly high among outdoor workers. South Asia has millions of bicycle rickshaw drivers, who use their muscles or battery power to pull hundreds of pounds of passengers and goods on modified bicycles. When manual rickshaw drivers rest to cool off, they reduce their already meager income. Heat stress not only threatens their livelihoods and thereby their right to an adequate standard of living but also their right to work, given that they have few employable skills other than manual labor. South Asia faces the greatest current and predicted loss in disability-adjusted life years due to heat stress, and heat stress is particularly strong in informal settlements. As such, the investigators plan to conduct this study in Dhaka, Bangladesh. The overall hypothesis is that driving a battery-powered rickshaw will reduce heat strain. The investigators will evaluate the impact of driving a battery-powered rickshaw on core temperature (primary outcome), telomere length, kidney function, heart rate, heart rate variability, sleep quality, self-reported thermal comfort, mental health, wellness, and fatigue (secondary outcomes).

ELIGIBILITY:
Inclusion Criteria:

* Reports driving a manual rickshaw at least five days per week for at least 8 hours per day for the past 12 months

Exclusion Criteria:

* Reports driving a battery-powered rickshaw in the past 12 months
* Has hypertension, as measured by our study staff
* Has diabetes, as measured by our staff
* Reports diagnosis with cardiovascular disease / chronic cardiac condition
* Reports diagnosis with respiratory disease / chronic respiratory condition

Min Age: 40 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Gender Based: Yes — Self-identify as a male. We will use this information about gender only as a proxy for sex, as we will not be assessing sex through chromosomal analysis.
Enrollment: 300 (Estimated)
Dates: Start 2025-06-01 (Estimated); Primary Completion 2025-10-31 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Core temperature | 0 (pre-intervention) and 2, 4, 6, 8, 10, 12, 14, 16 weeks post-intervention
  Minutes per day that core temperature is >40C, where fewer minutes per day is better

SECONDARY OUTCOMES:
Relative Leucocyte Telomere Length | 0 (pre-intervention) and 16 weeks post-intervention
  Change in Relative Leucocyte Telomere Length measured by PCR, where a smaller reduction in length is better
Kidney function | 0 (pre-intervention) and 2, 4, 6, 8, 10, 12, 14, 16 weeks post-intervention
  kidney function, as measured by a the neutrophil gelatinase-associated lipocalin (NGAL) value in urine samples, where a lower score is better
Heart rate | 0 (pre-intervention) and 2, 4, 6, 8, 10, 12, 14, 16 weeks post-intervention
  resting heart rate (bpm), where a lower heart rate is better
Heart rate variability | 0 (pre-intervention) and 2, 4, 6, 8, 10, 12, 14, 16 weeks post-intervention
  resting heart rate (bpm) variability, where higher variability is better
Sleep quality | 0 (pre-intervention) and 2, 4, 6, 8, 10, 12, 14, 16 weeks post-intervention
  Self-reported sleep quality and number of minutes in REM, as recorded by a fitness watch, where more minutes in REM is better

CONTACTS AND LOCATIONS:
Overall Officials: Laura Kwong, PhD, Principal Investigator — University of California, Berkeley

IPD SHARING:
Plan to Share IPD: Yes
We will post de-identified participant data on our OSF repository (https://osf.io/sd285/)
Supporting Information: Study Protocol, SAP, ICF, Analytic Code
Time Frame: We expect that data and code will become available by 1 Jan 2027